CLINICAL TRIAL: NCT00217529
Title: A Phase I-II Study of OSI-774 (Tarceva, Erlotinib) With Docetaxel/Carboplatin Followed by Maintenance Therapy With Tarceva as Treatment for Newly Diagnosed Stage III/IV Epithelial Ovarian Cancer, Primary Peritoneal or Fallopian Tube Cancer
Brief Title: Erlotinib, Docetaxel, and Carboplatin in Treating Patients With Newly Diagnosed Stage III or Stage IV Ovarian Epithelial, Primary Peritoneal Cavity, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Purpose: Treatment
Other Study IDs: PSOC 2001; PSOC-2001; AVENTIS-PSOC-2001; PSOC-IRB-5689; CDR0000441312 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; peritoneal cavity cancer; ovarian clear cell cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian undifferentiated adenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian serous cystadenocarcinoma; Brenner tumor; fallopian tube cancer; ovarian mixed epithelial carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — pegfilgrastim; Carboplatin; Docetaxel; Erlotinib Hydrochloride

INTERVENTIONS:
Biological: pegfilgrastim
Drug: carboplatin
Drug: docetaxel
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving erlotinib together with docetaxel and carboplatin may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of erlotinib when given together with docetaxel and carboplatin and to see how well they work in treating patients with newly diagnosed stage III or stage IV ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of erlotinib when administered in combination with docetaxel and carboplatin as front-line therapy in patients with newly diagnosed stage III or IV ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer.

Secondary

* Determine the toxicity of maintenance therapy with erlotinib when administered after front-line therapy in these patients.
* Determine the proportion of patients who are able to receive the full schedule of treatment courses.
* Determine the objective response rate in patients with measurable or evaluable disease treated with this regimen.
* Determine the progression-free and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of erlotinib.

* Front-line therapy: Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1, pegfilgrastim subcutaneously on day 2, and oral erlotinib once daily on days 3-16. Treatment repeats every 21 days for up to 6 courses.

Cohorts of 5 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 5 patients experience dose-limiting toxicity.

* Maintenance therapy: Beginning 3-4 weeks after the completion of front-line therapy, patients with stable or responding disease receive oral erlotinib once daily for up to 12 months.

After completion of study treatment, patients are followed every 6 months for 1 year and then periodically thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer

  * Stage III or IV disease
* The following histologic epithelial cell types are allowed:

  * Serous adenocarcinoma
  * Mucinous adenocarcinoma
  * Clear cell adenocarcinoma
  * Endometrioid adenocarcinoma
  * Mixed epithelial carcinoma
  * Undifferentiated carcinoma
  * Transitional cell carcinoma
  * Malignant Brenner tumor
  * Adenocarcinoma not otherwise specified
* Must have undergone appropriate surgery for ovarian epithelial, primary peritoneal cavity, or fallopian tube cancer within the past 6 weeks
* No borderline ovarian tumor of low malignant potential

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* Meets 1 of the following criteria:

  * Alkaline phosphatase (AP) normal AND AST or ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal
* No hepatic disease that would preclude study participation

Renal

* Creatinine ≤ 2.0 mg/dL
* Creatinine clearance > 50 mL/min
* No renal disease that would preclude study participation

Cardiovascular

* LVEF ≥ lower limit of normal*
* No poorly controlled arrhythmia
* No unstable coronary artery disease
* No myocardial infarction within the past year NOTE: *LVEF evaluation performed only on patients requiring it

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No peripheral neuropathy ≥ grade 2
* No other nonmalignant systemic disease that would preclude study participation
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No medical, social, or psychosocial factor that would preclude study participation
* No psychiatric or addictive disorder that would preclude giving informed consent
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix or breast

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for this malignancy

Chemotherapy

* No prior chemotherapy for this malignancy

Endocrine therapy

* No prior hormonal therapy for this malignancy

Radiotherapy

* No prior radiotherapy for this malignancy

Surgery

* See Disease Characteristics
* No planned interval cytoreductive surgery

  * Second-look surgery allowed

Other

* More than 1 year since prior experimental or investigational therapy
* No concurrent therapeutic anticoagulation with warfarin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of erlotinib

SECONDARY OUTCOMES:
Toxicity of maintenance therapy
Proportion of patients who receive the full schedule of treatment courses
Response rate
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Study Chair — Fred Hutchinson Cancer Center; Dan Veljovich, MD, Study Chair — Pacific Gynecology Specialists
Locations (3):
- United States (3):
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington